CLINICAL TRIAL: NCT02286349
Title: Effects of Noninvasive Brain Stimulation on Attentional Performance of Adults With Symptomatology of Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Non Invasive Brain Stimulation Effects on Attentional Performance in ADHD Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, PHD, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: ADHD_ brain stimulation_adults
Record Dates: First submitted 2014-11-04; First posted 2014-11-07 (Estimated); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Attention Deficit/Hyperactivity Disorder
Keywords: Neuromodulation Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Real rTMS group (Experimental): Submitted to 20 minutes of neuropsychological assessment (on average) + 5 blocks of real stimulation intensity of 10 Hz, each block containing 15 series of repetitive transcranial magnetic stimulation with 1 second duration and presenting interval of 10 seconds between sets + 20 minutes of neuropsychological reassessment (on average).
  Interventions: Device: Transcranial magnetic stimulation (Neurosoft®)
- Sham rTMS group (Sham Comparator): Submitted to 20 minutes of neuropsychological assessment (on average) + 5 stimulation sham blocks, each block containing 15 series of repetitive transcranial magnetic stimulation with 1 second duration and presenting interval of 10 seconds between sets + 20 minutes of neuropsychological reassessment (on average)
  Interventions: Device: Transcranial magnetic stimulation (Neurosoft®)
- Real tDCS group (Experimental): Submitted to 20 minutes of neuropsychological assessment (on average) + 10 minutes of real anodal transcranial direct current stimulation with intensity of 1 mA + 20 minutes of neuropsychological reassessment (on average).
  Interventions: Device: Transcranial direct current stimulation (Soterix, USA)
- Sham tDCS group (Sham Comparator): Submitted to 20 minutes of neuropsychological assessment (on average) + 10 minutes of sham transcranial direct current stimulation + 20 minutes of neuropsychological reassessment (on average)
  Interventions: Device: Transcranial direct current stimulation (Soterix, USA)

INTERVENTIONS:
Device: Transcranial magnetic stimulation (Neurosoft®) — Repetitive transcranial magnetic stimulation
  Arms: Real rTMS group; Sham rTMS group
Device: Transcranial direct current stimulation (Soterix, USA) — Transcranial direct current stimulation
  Arms: Real tDCS group; Sham tDCS group

SUMMARY:
This study aims to evaluate the effect of noninvasive brain stimulation in adults with ADHD symptomatology compared them with healthy adults. For this, volunteers will allocate into two groups (experimental and control), will pass through session two types of transcranial stimulation: Repetitive Transcranial MagneticsStimulation (rTMS) and transcranial direct current stimulation (tDCS); considering two session types (real and sham). Attentional assessment will be carried out through specific neurocognitive tests applied before and after each session of stimulation

DETAILED DESCRIPTION:
The sample will be divided into four groups: (i) Experimental tDCS; (ii) Experimental rTMS; (iii) tDCS control; and rTMS control. The experimental groups consisted of subjects with ADHD symptomatology. Control groups were formed by healthy individuals.

The subject will be considered healthy when there was no diagnosis of any DSM-IV psychiatric disorder and had symptoms with ADHD when there were frequent presence of at least six symptoms of inattention and / or symptoms of hyperactivity/impulsivity described by the Adult Self Report Scale (ASRS), a reliable tool for diagnosis of attention deficit / hyperactivity and validated for the Brazilian population.

Both groups underwent two sessions of cortical stimulation: real (rTMS or tDCS) and sham. The order of sessions will be randomized and there will be a minimum interval of at last one week between sessions.

Experimental Sessions

Repetitive Transcranial Magnetic Stimulation (rTMS) With the individual seated comfortable, rTMS will be applied through a magnetic stimulator (Neurosoft®) using a figure-8 coil, positioned on the scalp at an angle of 45 degrees from the midline and pointing toward the anterior region of the skull.

The area stimulated will be the left dorsolateral prefrontal cortex (DLPFC). Before applying rTMS over the DLPFC will be necessary to map the area of the representation of the FID by applying single pulses to measure the motor evoked potential (MEP) and resting motor threshold (RMT). The intensity adopted in real rTMS session will be 80% of the RMT. rTMS will be applied in just one session divided in to 5 blocks of stimulation. Each block will be separated by 5 minutes intervals. In each block 15 rTMS series of 1-second duration at 10 Hz frequency were applied. The interval between sets will be 10 seconds. The sham stimulation will be applied with the same settings real rTMS, but the coil will be not coupled to the magnetic stimulator, so the individual will be not able to differentiate the real session of sham.

Transcranial Direct Current Stimulation (tDCS) Individuals will be instructed to sit in a chair and get a comfortable position. The continuous electrical current will be applied through a microcurrent stimulator (Soterix, USA). The surface electrodes used in all sessions of this study have dimensions of 5x7cm (35 cm2), were composed of electrically conductive rubber and wrapped in sponges soaked in saline.

For the application of tDCS, the anode will be positioned on DLPFC and cathode in the contralateral supraorbital region. Parameters of intensity and stimulation duration of the current used were previously established in humans: intensity 1mA and duration of 10 minutes. In sham stimulation, sessions will use the same procedures of real tDCS application, however the stimulation device will be switched off five seconds after the start.

Outcome measures - The subjects will be submitted an evaluation before (t0) the application of non-invasive cortical stimulation (active and sham) and immediately after (t1). These assessments consisted of neurocognitive tests that assess cognitive function and attention span of the patients. The tests will be applied (i) Trail Making Test (part A and B); (ii) digit span (forward and reverse order); (iii) digit symbol; (iv) C; (v) D2. Thus, the following items were assessed: (i) attentional focus (digit symbol, AC and trail making-part A); (ii) maintaining the attentional focus (D2 test); (iii) attentional span (digit span forward); (iv) the ability of mental manipulation (digit span backward and trail making test- part B); (v) ability to resist interference (D2 test).

Neuropsychological assessment will be performed by a neuropsychology, blind to the type of experimental session (rTMS / or active tDCS / sham) to which the subject was submitted.

ELIGIBILITY:
Inclusion Criteria:

Experimental group Punctuate 6 items or more (in the "frequently" and / or "quite often" on the Adult Self Report Scale (ASRS-18).

* Control group Punctuate fewer than six items (in the "frequently" and / or "quite often" on Adult Self Report Scale (ASRS-18) Not exhibit symptoms of other disorders measured by the Mini International Neuropsychiatric Interview (M.I.N.I).

Exclusion Criteria:

* epilepsy;
* neurosurgery (including implant metal clips);
* head trauma;
* implantation of a pacemaker;
* current use of epileptogenic drugs;
* uncontrolled severe organic disease.
* pregnancy.
* current use of psychostimulant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Digit Span (forward and backward) | The test will be administered before and after each stimulation session for all groups involved in the research. The stimulation sessions present an interval of one week. The whole rTMS session will last 30 minutes and the tDCS session of 10 minutes. The
  The digit span forward contains eight items of sequence numbers that should be recalled in direct order after reading the examiner and digit span backward contains seven items of sequences of numbers that should be recalled in reverse order. Both are interrupted when two sequences of the same item number is wrong.

SECONDARY OUTCOMES:
D2 test | The test will be administered before and after each stimulation session for all groups involved in the research. The stimulation sessions present an interval of one week. The whole rTMS session will last 30 minutes and the tDCS session of 10 minutes. The
  Characterized as a test of concentrated visual attention and in the broadest sense, the ability to concentrate. It consists of 14 lines, the subjects must identify and scratch at each line the letters "d" having two lines, having a time limit of 20 seconds to complete each line
Trail Making Test (A and B) | The test will be administered before and after each stimulation session for all groups involved in the research. The stimulation sessions present an interval of one week. The whole rTMS session will last 30 minutes and the tDCS session of 10 minutes. The
  Participants are required to draw a line connecting numbered circles in a sequential order in part A. In part B the same task is performed, however, the participant must connect numbered and lettered circles in alternating sequential-alphabetical order. The TMT is presented as a measure of attention, processing speed and mental flexibility.
Digit Symbol Modality Test | The test will be administered before and after each stimulation session for all groups involved in the research. The stimulation sessions present an interval of one week. The whole rTMS session will last 30 minutes and the tDCS session of 10 minutes. The
  The SDMT requires individuals to identify nine different symbols corresponding to the numbers 1 through 9, and to practice writing the correct number under the corresponding symbol. Then they manually fill the blank space under each symbol with the corresponding number. It is a test used to investigate divided attention, visual tracking and motor processing speed.
AC Test | The test will be administered before and after each stimulation session for all groups involved in the research. The stimulation sessions present an interval of one week. The whole rTMS session will last 30 minutes and the tDCS session of 10 minutes. The
  The test aims at maintaining concentrated attention at work. The test consists of 21 lines, each having 21 symbols so that each line should be canceled whenever 7 symbols. The stimuli that must be canceled are found in a rectangle on top of the sheet

CONTACTS AND LOCATIONS:
Overall Officials: Kátia Monte-Silva, PHD, Principal Investigator — Applied Neuroscience Laboratory, Universidade Federal de Pernambuco